CLINICAL TRIAL: NCT00169793
Title: Nephrolithiasis and Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 05-076
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Obesity; Nephrolithiasis
Keywords: Obesity; Nephrolithiasis
MeSH Terms: conditions — Obesity; Nephrolithiasis | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other)
  Interventions: Other: evaluation of kidney stone risk after bariatric surgery; Other: Evaluate risk of kidney stones after bariatric surgery

INTERVENTIONS:
Other: evaluation of kidney stone risk after bariatric surgery — 24 hour urine collections done pre and post surgery
  Other Names: observation
Other: Evaluate risk of kidney stones after bariatric surgery — 24 hour urine collections are done before and after surgery
  Other Names: observation

SUMMARY:
Test the hypothesis that the new bariatric surgical procedures (BSP) increase stone risk, and will result in an increased incidence and prevalence of stone disease; the purpose is to determine if BSP patients require special management for stone prevention. This study does not include the bariatric surgery but enrolls subjects who are already scheduled for surgery with an affiliated surgeon. The study procedure is to collect 24 hour urines pre-and post surgically to evaluate the risk of kidney stone procedure after surgery.

DETAILED DESCRIPTION:
Surgical therapy for the morbidly obese began when the jejunocolic anastomosis procedure was performed in 1956 but was modified to a jejunoileal technique years later after intolerable metabolic complications ensued.1, 2 In 1969, Payne recommended that the end to side jejunal-ileal bypass (JIB) procedure which preserved 37cm of jejunum and 10cm of ileum should replace the jejunocolic bypass.2 In 1970, Scott modified JIB by increasing the length of intestine used and by fashioning an end-to-end anastomosis between the jejunum and ileum3; this modified procedure soon became the preferred procedure for weight reduction. This foray into bariatric surgery was quickly embraced and JIB was widely adopted. However, in the mid to late 1970's, about 10 years after the first JIB was performed, concern developed regarding the long-term adverse effects of anemia, vitamin deficiencies, nephrolithiasis and ultimately even renal and liver failure.4-14 It was not until a number of patients had end organ failure that the full impact of the complications of JIB were recognized. Much of the complications stem from the malabsorptive component that results from JIB. As fat is malabsorbed, fat-soluble vitamins and calcium are saponified. Subsequently, nutrients are lost and an increased oxalate load is delivered to the large intestine as the calcium that would normally bind oxalate is lost with the malabsorbed fat. In addition, bile salts normally reabsorbed in the ileum are delivered to the colon, increasing the permeability of the colonic mucosa to oxalate. These factors result in increased uptake of oxalate in the large intestine. Oxalate, which cannot be metabolized by humans, is rapidly cleared by the kidney resulting in "intestinal" hyperoxaluria and calcium oxalate nephrolithiasis4-6, 12, 15 and nephrotoxicity.7, 10, 11, 13, 16 The probability of a severe renal complication after JIB was calculated to be about 21% at 5 years and increased to 37% at 15 years; there is also a 28.7% risk of nephrolithiasis at 15 years.13 It was not until 1980 that the Food and Drug Administration placed a moratorium on JIB for obesity surgery. Prior to that approximately 25,000 such procedures had been performed in the United States. A large number of these patients had the JIB reversed or succumbed to its complications.10 Those patients with the JIB intact remain at risk for complications such as cirrhosis, arthritis, urolithiasis, oxalate nephropathy, and bypass enteritis-of which only the latter three respond when the JIB is reversed.10 The lessons learned from this previous experience with bariatric surgical procedures must not be repeated. Although the cardiopulmonary risks of obesity are significant, the catastrophic long-term consequences that were unrecognized initially with JIB should not be forgotten. Many patients not only necessitated treatment for kidney stones but some have lost renal function requiring dialysis and transplantation from oxalate nephropathy.10, 11, 13 Currently, the Roux-en-Y bariatric procedure (REY) is the most widely utilized procedure for the surgical treatment of obesity. REY results in rapid weight loss17 compared to restrictive procedures16, 17, 18-20 but the long-term effects of the malabsorptive component of this operation on the risk of nephrolithiasis and renal loss is currently unknown. With REY, fat malabsorption is one of the primary mechanisms by which weight loss is accomplished and, therefore, intestinal hyperoxaluria, as occurs with JIB, is theoretically possible. Although the long-term metabolic consequences of REY have yet to be studied, some recent data from LithoLink is concerning. LithoLink Corporation, located in Chicago IL, is a clinical laboratory/disease management company that provides testing for kidney stone patients. Physicians from all across the United States refer stone patients to the LithoLink laboratory for evaluation. Patients collect 24-hour urine samples at home and then send them via overnight air express to LithoLink for analysis. As part of the disease management service, a medical history pertinent to kidney stones is obtained from each patient via phone interview. Since 1998, patients have specifically been asked if they have had weight reduction surgery and whether the surgery was JIB or bariatric, and the answers are coded into the database. The LithoLink database is the largest kidney stone database linking laboratory and clinical data in this country, and perhaps the world. As part of an IRB approved research protocol, LithoLink sought to ask the question whether modern bariatric procedures were associated with an increase in urine oxalate excretion. They found normal non-stone forming controls have a mean urinary oxalate excretion of 34.3mg/day while calcium oxalate stone formers from the same laboratory have a mean urinary oxalate excretion of 37.3mg/day. In contrast, the bariatric population, which includes both gastric banding (restrictive only) and REY (restrictive and malabsorptive) patients, was found to have a mean urinary oxalate excretion of 78.4mg/day (p<0.001 compared to both normal controls and stone formers). Figure 1 shows the comparison of urine oxalate excretion of bariatric surgery patients to that of routine stone formers. Note the significant right shift to higher oxalate excretion in the bariatric surgery patients (open triangles). Most laboratories consider a urinary oxalate excretion of >45mg/day to represent hyperoxaluria and primary hyperoxaluria (a rare inborn error of metabolism resulting in marked endogenous production of oxalate) is suspected when the level of urinary oxalate exceeds 100mg/day6. Given these definitions, the urine oxalate excretion in patients having undergone bariatric surgery is striking. Nearly 3/4 of the bariatric surgery cohort had urine oxalate levels above 45mg/day and about 1/4 had urinary oxalate levels in excess of 100mg/day. Calcium oxalate supersaturation (Figure 2), the chemical driving force for crystallization, is also dramatically elevated in bariatric surgery patients compared to routine stone formers (12.5 vs. 7.3, p<0.001), highlighting the extreme risk for stone formation and oxalate nephropathy in these patients. Finally, the data was analyzed to see if there was an increase in the number of bariatric surgery patients being referred for kidney stone evaluation. Since the number of new patients referred to Litholink each year is increasing, the data is presented as the number of new bariatric surgery patients per one thousand new stone patients per year. As can be seen in Figure 3, there is a significant upward trend of bariatric surgery patients with kidney stones (r2= 0.86 for the linear regression, p=0.01). This rise in bariatric surgery patients with kidney stones parallels, but lags by several years, the rise in the number of bariatric surgeries in the United States (Figure 3). Although bariatric procedures such as REY are performed with the assumption that the resultant physiologic perturbations should be less severe than with JIB, our preliminary data suggests that these contemporary bariatric surgical procedures result in urinary oxalate levels comparable to that reported after JIB with the now well-known long-term adverse sequela vis-à-vis nephrolithiasis and oxalate nephropathy.

Because Clarian, as well as many other medical institutions, is undertaking a large endeavor to become a center of excellence in bariatric surgical treatment, the risk of stone formation and renal disease in these patients should be carefully examined. It is hoped that early recognition of adverse metabolic alterations will allow the patient and physician to rapidly treat and even prevent some complications. Loss of renal function, as with the previous experience with JIB, is much too late a phase in the consequences of hyperoxaluria for the identification of such problems associated with bariatric surgery. Patients can also be adequately counseled if they have a prior history of stone disease regarding the relative risks of the various bariatric surgical procedures. As obesity is currently an important national health issue, the examination of the surgical treatment for obesity and the consequences of these procedures is timely. Scrutiny of the risks of bariatric surgery will benefit both patient and surgeon in identify and preventing renal complications that may arise.

ELIGIBILITY:
Inclusion Criteria:

* Already scheduled to undergo bariatric surgery with a Clarian affiliated surgeon in Indianapolis, IN
* Over the age of 18
* Able to give informed consent
* Able to comply with 24 hour urine collections at specified times

Exclusion Criteria:

* Not scheduled for bariatric surgery
* Bariatric surgery to be done by a non-Clarian affiliated surgeon
* Unable to give informed consent
* Unwilling/unable to comply with 24 hour urine collections at specified times

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-08; Primary Completion 2009-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To quantify the prevalence of stone disease among patients at the Clarian Hospitals who have had BSP between 3 and 3.5 years previously. | In the next two years

SECONDARY OUTCOMES:
To identify clinical and laboratory risk factors for incident nephrolithiasis following bariatric surgery. | In the next two years

CONTACTS AND LOCATIONS:
Overall Officials: James E. Lingeman, MD, Principal Investigator — Methodist Urology, LLC
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States